CLINICAL TRIAL: NCT03395561
Title: the Evaluation of Green Coffee Extract Supplementation on Adropin, Irisin, Vaspine,Systemic Inflammation and Oxidative Stress in Breast Cancer Survivors
Brief Title: Effects of Green Coffee Extract Supplementation on Adropin, Irisin, Vaspine,Systemic Inflammation and Oxidative Stress in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 811
Record Dates: First submitted 2017-12-26; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer Survivors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- green coffe (Active Comparator): 2 capsuls of green coffe
  Interventions: Dietary Supplement: green coffee
- control (Placebo Comparator): 2 capsuls
  Interventions: Other: control

INTERVENTIONS:
Dietary Supplement: green coffee — 2 capsuls
  Arms: green coffe
Other: control — 2 capsuls
  Arms: control

SUMMARY:
To study the effects of green coffee supplement on adropin, irisin, vaspine, systemic inflammation and oxidative stress in breast cancer survivors.50 breast cancer survivors who their treatment is over and referred to follow breast cancer clinic with will be randomly allocated to receive placebos or 2 capsules green coffe for 12 weeks; both groups will be advised to adherence the investigators' diet and exercise program too. At the first and the end of the intervention, adropin, irisin, vaspine, systemic inflammation and oxidative stress will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) between 25-40 treatment is over

Exclusion Criteria:

* Taking any kind of supplement for weight reduction
* pregnancy or lactation
* Professional athletes

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-11 (Estimated); Primary Completion 2019-01-11 (Estimated); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Tumor necrosis factor alpha | 12 weeks
  assessed by ELISA
Interleukin 6 | 12 weeks
  assessed by ELISA

SECONDARY OUTCOMES:
body mass index | 12 weeks
  The body mass index (BMI) or Quetelet index is a value derived from the mass (weight) and height of an individual. The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran